CLINICAL TRIAL: NCT01836380
Title: Effects of Swimming Exercise and Cycling Exercise Interventions on Vascular Function, Inflammation and Pain in Middle-aged and Older Adults With Osteoarthritis.
Brief Title: Regular Swimming, Vascular Function, and Arthritis
Acronym: OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOA26752611
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Swimming Training (Experimental): The swimming training will be performed at two swimming pools on the campus of The University of Texas at Austin (University Aquatic Center or Gregory Gym pool). In the first 2-3 weeks a swimming instructor will provide personalized skill feedback to the subjects in the swim training group. Subjects will swim 15-20 minutes/day at a relatively low intensity of exercise while they receive swimming skill instructions. As their overall level of fitness and exercise skill improve, the intensity and duration of exercise will increase to 40-45 minutes/day at a moderate intensity of 70-75% of maximal heart rate. Exercise training will be performed three days per week.
  Interventions: Behavioral: Exercise Training
- Cycling Training (Experimental): The cycling training will be conducted in the newly-constructed Exercise Training Intervention Core-Laboratory in the Department of Kinesiology and Health Education on the University of Texas campus. In the first 2-3 weeks a cycling instructor will provide personalized skill feedback to the subjects in the cycle training group. Subjects will cycle 15-20 minutes/day at a relatively low intensity of exercise while they receive cycling skill instructions. As their overall level of fitness and exercise skill improve, the intensity and duration of exercise will increase to 40-45 minutes/day at a moderate intensity of 70-75% of maximal heart rate. Exercise training will be performed three days per week.
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training

SUMMARY:
Hypothesis #1: The investigators hypothesize that both swimming training and cycling training will demonstrate significant improvements in endothelium-mediated vasodilation and central artery compliance in this population and that there will be no difference in the magnitude of increases between the water-based and land-based exercise interventions.

Hypothesis #2: The investigators hypothesize that the improvements in endothelium-dependent vasodilation and arterial compliance in response to exercise training interventions will be related to the corresponding reductions in inflammatory biomarkers.

Hypothesis #3: The investigators hypothesize that both swimming exercise and cycling exercise will improve functional capacities and disease progression in middle-aged and older adults with osteoarthritis.

DETAILED DESCRIPTION:
Middle-aged and older men and women (40-90 years old) of all races and ethnic backgrounds will serve as subjects after obtaining their written, informed consent. All the subjects will have a radiological diagnosis of osteoarthritis according to American College of Rheumatology criteria.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects will have a radiological diagnosis of osteoarthritis according to American College of Rheumatology criteria
* Subjects will be sedentary (i.e., no regular physical activity for at least the prior 1 year)

Exclusion Criteria:

* Subjects with significant intima thickening,
* plaque formation, and/or characteristics of atherosclerosis.
* unstable cardiac or pulmonary diseases.
* joint replacement surgery in the previous year.
* intraarticular injection nor systemic steroids within previous 3 months.
* severe disabling co-morbidity that disallows receiving exercise therapy.
* excess alcohol use (>21 drinks/week).
* unwillingness to perform exercise.
* fear of water.
* mental incapability

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Central Arterial Compliance | three months
  Central Arterial Compliance: Common carotid artery diameter will be measured from the images derived from an ultrasound machine (Philips HDI-5000, Bothel, WA) equipped with a high-resolution linear-array transducer as previously described. A longitudinal image of the cephalic portion of the common carotid artery will be acquired 1-2 cm proximal to the carotid bulb with the transducer placed at 90 degrees to the vessel. The images will be analyzed with Vascular Tools 5 image analyses software. Similarly, intima-media thickness will be measured at end diastole as previously described. The combination of ultrasound imaging of a common carotid artery with simultaneous tonometric-obtained arterial pressure waveforms from the contralateral artery permits noninvasive determination of carotid artery compliance. Arterial compliance is a function of the increase in arterial pressure and a corresponding increase in cross-sectional area.
Inflammatory Markers | three months
  Fasted state, venous blood samples will be obtained to assess biological markers of inflammation. Serum C-reactive protein (CRP) will be assayed using ELISA (Alpha Diagnostics; San Antonio, TX). Inflammatory cytokines including Interleukin-6 (IL-6), TNF-α, and soluble receptor 1 (sTNFR1) will be analyzed from serum samples using a multiplex assay system (Bioplex, BioRad; Hercules, CA)
Flow-Mediated Dilatation | three months
  Flow-Mediated Dilatation is a non-invasive method to assess vascular endothelial function as previously described. Brachial artery diameters and blood flow velocity will be measured from images derived from a Doppler ultrasound machine equipped with a high-resolution linear array transducer. A longitudinal image of the brachial artery will be acquired 5-10 cm proximal to the antecubital fossa. A blood pressure cuff will be placed on the forearm 3-5 cm distal to the antecubital fossa. The cuff will be inflated to 100 mmHg above resting systolic blood pressure for 5 minutes. After cuff deflation, ultrasound-derived measurements of the brachial artery diameters and blood velocity will be taken for 3 minutes. FMD will be calculated as a percent increase in brachial artery diameter at the post-blood flow occlusion compared with the pre-blood flow occlusion.

SECONDARY OUTCOMES:
Mobility | three month
  Six-minute walk distance will be used for a measure of mobility and functional status. Participants will be instructed to walk as far as possible on a flat, indoor surface.
Muscular Strength | three months
  Bilateral isometric quadriceps strength will be measured in order to evaluate the impact of exercise intervention on lower body strength. Grip strength will also be measured using standard grip strength dynamometer.
Body Mass and Composition | three months
  Body mass will be measured to the nearest 0.1 kg with a physicians' balance scale (SECA, Hamburg, Germany). Body composition will be determined using dual-energy x-ray absorptiometry (DEXA)(GE Lunar Radiation, Madison, WI).
Self-Reported Physical Function and Pain | three months
  A self-report questionnaire, the Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) will be used to assess the degree of difficulty in performing activities of daily living. It consists of 17 questions that generate a summary score ranging from 0-68, with higher scores indicating increased disease severity.
Health-Related Quality of Life | three months
  Participants will complete the Short Form Health Survey (SF-36) questionnaire. The SF-36 survey consists of two subscales including physical health and mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Alkatan M, Baker JR, Machin DR, Park W, Akkari AS, Pasha EP, Tanaka H. Improved Function and Reduced Pain after Swimming and Cycling Training in Patients with Osteoarthritis. J Rheumatol. 2016 Mar;43(3):666-72. doi: 10.3899/jrheum.151110. Epub 2016 Jan 15. PMID 26773104
- [Derived] Alkatan M, Machin DR, Baker JR, Akkari AS, Park W, Tanaka H. Effects of Swimming and Cycling Exercise Intervention on Vascular Function in Patients With Osteoarthritis. Am J Cardiol. 2016 Jan 1;117(1):141-5. doi: 10.1016/j.amjcard.2015.10.017. Epub 2015 Oct 22. PMID 26541906